CLINICAL TRIAL: NCT01298778
Title: Improving Pain Relief For Those Who Need It Most After Cesarean Delivery
Brief Title: High Pain Intervention in Cesarean Sections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00012376
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Results first posted 2017-06-09 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Other Chronic Postoperative Pain
Keywords: chronic pain post delivery; postpartum depression; tailored pain management
MeSH Terms: conditions — Depression, Postpartum | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Placebo Comparator): Spinal consists of duramorph 150 mcg combined with fentanyl and bupivacaine in conjunction with placebo capsules 2 PO q 6 hrs x 4 doses in first 24 hrs postop. Ibuprofen given as standard of care.
  Interventions: Drug: Duramorph 150
- Acetaminophen and increased dose of Duramorph (Active Comparator): Spinal consists of duramorph 300 mcg combined with fentanyl and bupivacaine in conjunction with Acetaminophen 1 Gm PO q 6 hrs x 4 doses in first 24 hrs postop. Ibuprofen given as standard of care.
  Interventions: Drug: Acetaminophen; Drug: Duramorph 300

INTERVENTIONS:
Drug: Duramorph 150 — Duramorph 150 mcg x 1 dose spinally + placebo capsules 2 PO q 6 hrs first 24 hrs postop x 4 doses
  Arms: Standard of care
Drug: Acetaminophen — Duramorph 300 mcg spinally + acetaminophen 1 GM q 6 hrs first 24 hrs postop x 4 doses
  Arms: Acetaminophen and increased dose of Duramorph
Drug: Duramorph 300 — Duramorph 300 mcg spinally + acetaminophen 1 GM q 6 hrs first 24 hrs postop x 4 doses
  Arms: Acetaminophen and increased dose of Duramorph

SUMMARY:
In previous studies the investigators have seen that the severity of pain one day after cesarean delivery can predict the presence of pain and depression 2 months later. The investigators believe those at risk for severe acute post-partum pain can be identified, and medical interventions can be tailored to manage postoperative pain more effectively.

DETAILED DESCRIPTION:
This study is randomizing patients into 2 different groups and seeing if by altering our pain management with this group of patients their acute 24 hour evoked pain is less than anticipated; and the incidence of persistent pain and depression when contacted 2 months after delivery is decreased. This study is designed to see if these additional interventions would prove effective for patients at risk of having high pain level after cesarean surgery.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean section
* age >/= 18 years old
* not allergic proposed study medications
* predicted to experience high pain postop based on preoperative evaluation

Exclusion Criteria:

* allergy to study medications
* known hepatic disease
* weight > 300 lbs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter H. Pan, MD, MSEE, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Forsyth Medical Center-Sara Lee Center for Women's Health, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were approached during the pre-anesthesia evaluation regarding their interest in the study. Once consent was signed, subjects completed their pre-surgery questionnaires. On the day of surgery, I/E criteria were re-reviewed for confirmed enrollment for study.A total of 74 were consented with 69 randomized, with 60 completing the study.
Groups:
- Standard of Care: Spinal consists of duramorph 150 mcg combined with fentanyl and bupivacaine in conjunction with placebo capsules 2 PO q 6 hrs x 4 doses in first 24 hrs postop. Ibuprofen given as standard of care.
  Duramorph: Duramorph 150 mcg x 1 dose spinally + placebo capsules 2 PO q 6 hrs first 24 hrs postop x 4 doses
Period: Overall Study
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Started | 33 | 36
Completed | 30 | 30
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 2 | 3
Not completed — Incorrect use of VAS | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — not meet inclusion/exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants] — years of age at time of consent
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 30 | 30 | 60
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 30 | 60
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
Height-cm [Mean (Standard Deviation); unit: cm] | 163 (6) | 164 (6) | 163.3 (6)
Weight-kg [Mean (Standard Deviation); unit: kg] | 88 (17) | 92 (19) | 89.7 (17.7)
Gestational Age-weeks [Mean (Standard Deviation); unit: weeks gestation] | 39 (0.3) | 39 (0.7) | 39 (0.5)
Parity [Mean (Full Range); unit: number previous deliveries] | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 2]
Previous Cesarean Section [Count of Participants; unit: Participants] — Number of subjects out of the total subjects per group that had experienced a previous CS Delivery
  Participants | 27 | 24 | 51
ASA class [Median (Full Range); unit: units on a scale] — American Society Anesthesiology classification of 1 (healthy), 2, 3, or 4 (most severely ill)
  units on a scale | 2 [1 to 4] | 2 [1 to 4] | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Severity of Acute Pain
Description: to determine whether an intervention in women predicted to experience severe pain after cesarean delivery reduces acute post-delivery pain (24 hour evoked pain post delivery). The scale utilized was a 100mm sliding VAS, where 0mm=no pain up to 100mm-worst pain imaginable.
Time Frame: 24 hour
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
mm | 46 (25) | 31 (17)
Statistical Analysis 1: Comparison: Acetaminophen and Increased Dose of Duramorph; acute pain scores with movement at 24 hours; Test type: Superiority or Other; p = 0.05, t-test, 2 sided

2. Secondary Outcome: Incidence of Persistent Pain
Description: to determine whether an intervention in women predicted to experience severe pain after cesarean delivery reduces persistent pain up to 2 months post delivery.
Time Frame: 2 months
Measure: Number; unit: percentage of participants
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
percentage of participants | 13 | 10

3. Secondary Outcome: Pain
Description: resting pain, worst pain
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: units on a scale, 0 -none, 100-worst
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
units on a scale, 0 -none, 100-worst
  resting pain score over 24 hrs | 19 [0 to 33] | 4 [0 to 10]
  worst pain score over 24 hrs | 69 [49 to 77] | 62 [42 to 70]

4. Secondary Outcome: Analgesic Consumption
Description: total amount of analgesic consumption
Time Frame: 24 hour
Measure: Median (Inter-Quartile Range); unit: mg
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
mg
  IV PCA morphine | 15 [11 to 32] | 15 [11 to 29]
  total 24 hr opioid use | 21 [11 to 37] | 15 [13 to 33]

5. Secondary Outcome: Incidence of Depression
Description: to determine whether an intervention in women predicted to experience severe pain after cesarean delivery reduces postpartum depression up to 2 months post delivery.
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
Participants | 3 | 4

6. Secondary Outcome: Average Pain Over 24 Hours
Time Frame: 24 hours
Population: VAS pain score of 0=no pain at all up to 100 being worst pain imaginable.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
units on a scale | 37 (19) | 23 (14)

7. Other Pre Specified Outcome: Pruritus
Description: side effects-percentage of subjects requiring treatment
Time Frame: 24 hours
Population: percentage of patients with pruritis requiring treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
Participants | 15 | 21

8. Other Pre Specified Outcome: Emetic Symptoms
Description: side effect potential with the increased dose of duramorph-percentage experiencing such symptoms
Time Frame: 24hours
Population: percentage of patients reporting emetic symptoms requiring treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Number analyzed (Participants) | 30 | 30
Participants | 16 | 18

ADVERSE EVENTS:
Time Frame: Participants were followed at 24 hours postoperatively and for 8 weeks postpartum.
Description: Outcome measures for incidence of pruritis and emetic symptoms have been reported in the arms section as those were expected outcomes that could be measurable.
  These are all anticipated events for such surgery patients and do not exceed the normal frequency threshold; therefore they were not considered adverse events.
Arm/Group | Standard of Care | Acetaminophen and Increased Dose of Duramorph
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes